CLINICAL TRIAL: NCT01204151
Title: Evaluating a Brief Intensive Intervention for Individuals With Fragile X Syndrome
Brief Title: Teaching Math Skills to Individuals With Fragile X Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Hall, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SU-09132010-6849
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Developmental Disabilities; Fragile X Syndrome
MeSH Terms: conditions — Developmental Disabilities; Fragile X Syndrome

ARMS (1):
- Math intervention (Experimental)
  Interventions: Behavioral: discrete-trial training

INTERVENTIONS:
Behavioral: discrete-trial training

SUMMARY:
Children with FXS are predisposed to manifesting a particular profile of intellectual strengths and weaknesses, including specific deficits in math, visual-spatial skills, executive functioning, and social skills. Until now, intensive behavioral interventions have not been targeted to syndrome-specific weaknesses. In the present study we will develop and evaluate behavioral strategies to aid skill acquisition in children with FXS.

DETAILED DESCRIPTION:
There are no experimental data of skill acquisition using matching-to-sample techniques (or any other specific cognitive intervention) conducted with individuals with FXS. Further, no studies have been conducted to examine the possible underlying or mediating brain processes involved during matching-to-sample skill acquisition in children with FXS or any other neurodevelopmental disorder.

Previous pilot data have indicated that the computerized match-to-sample procedure, even when conducted in time-limited sessions, may significantly help individuals with FXS learn new skills. We plan to utilize brain imaging methodology to compare functional connectivity networks for those who pass and those who fail the equivalence test. 30 subjects with FXS and 30 control subjects with idiopathic developmental disability will be enrolled in the study. All subjects will be enrolled at Stanford.

ELIGIBILITY:
Inclusion Criteria:

* (a) 10 to 23 years of age (this age range was chosen to maximize the probability that subjects will cooperate with the imaging procedures as well as benefit from the interventions),
* (b) in good physical health,
* (c) able to participate in the imaging component of the project,
* (d) IQ between 50 and 80. We have found that individuals with IQ's less than 50 points are generally unable to comply with the scanning procedures.
* (e) diagnosis of FXS (for FXS group) and non-specific developmental disorder (for control group).

Exclusion Criteria:

Exclusion criteria include

* contraindications for MRI (e.g., pacemaker, braces),
* the presence of neurological or sensory problems not associated with the conditions of interest (e.g., head trauma, blindness), or inability to discontinue psychotropic medication for 4 weeks prior to the scan.
* Additional exclusion criteria for the control group include the presence of any known identifiable syndrome (e.g., fragile X syndrome, Down syndrome, Prader-Willi syndrome, Turner syndrome, PKU, fetal alcohol syndrome, Williams syndrome).

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percent correct | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hall, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States